CLINICAL TRIAL: NCT05604079
Title: Feasibility Assessment of the Electrolarynx for Enabling Communication in the
Brief Title: Electrolarynx for Enabling Communication in the CHrOnically Critically Ill (EECCHO)
Acronym: EECCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Garron Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TorontoEGH
Record Dates: First submitted 2015-01-05; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-05

CONDITIONS: Communication
Keywords: communication; mechanical ventilation; weaning
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrolarynx (Experimental): In this single arm study, all participants will receive training in the Electrolarynx
  Interventions: Device: Electrolarynx

INTERVENTIONS:
Device: Electrolarynx — The device transmits electronic sound source vibrations through soft tissue, either the neck at the level of the glottis, or less commonly the check. Speech is created through movements of articulators including the lips, tongue and jaw.

SUMMARY:
All critically ill patients receiving mechanical ventilation experience a period of inability to speak due to the need for cuffed endotracheal or tracheostomy tubes. Consequences of the inability to speak include: significant emotional distress; unrecognized pain; sleeplessness; increased use of restraints, self-extubation and line removal, as well as injury to self and healthcare professionals. Communication methods such as word mouthing, gesticulating, and writing may be ineffective and result in frustration. Recent technological innovations include communication boards and electronic speech generating devices however these require fine motor skills and coordination which may not be intact in the chronically critically ill. The Electrolarynx was recently shown to be effective in establishing communication in a case study of an intubated patient. Despite the well-recognized deleterious consequences of speech incapacity, few studies have evaluated communication strategies in the critically ill and no published study has evaluated the Electrolarynx in this patient population.

In this study, the investigators aim to assess the feasibility and patient acceptability of establishing speech with an Electrolarynx for intubated or tracheostomized patients experiencing difficult weaning and unable to tolerate cuff deflation. Feasibility will be determined by the proportion of participants able to produce intelligible and comprehensible speech. The investigators will also collect data on consent rates, reasons for refusal, the proportion of eligible patients and the time required for research procedures to inform future studies. The investigators will provide participants with a maximum of five Electrolarynx training sessions. On completion the investigators will measure speech intelligibility, comprehensibility, and patient acceptability using the Assessment of Intelligibility of Dysarthric Speech and the Ease of Communication scale. Satisfaction with communication and anxiety will be measured before and after Electrolarynx training. To the investigators' knowledge, this study will be the first to rigorously evaluate, using previously validated measures, the feasibility of the Electrolarynx for establishing communication for mechanically ventilated patients.

DETAILED DESCRIPTION:
Despite the well-recognized deleterious consequences of speech incapacity, few studies have evaluated communication strategies for patients unable to tolerate cuff deflation. Despite the aforementioned case reports, no studies report the feasibility of the Electrolarynx in restoring communication. Communication impairment during hospitalization has implications for the quality and safety of care as it is a modifiable risk factor for adverse events. This has led to accreditation organizations mandating reasonable efforts to establish alternative communication strategies for patients unable to speak. For chronically critically ill (CCI) patients, inability to speak increases anxiety, decreases a sense of control, and impairs meaningful patient involvement in decision making. Anxiety can exacerbate pain, which is known to impede ventilator weaning. Therefore it is likely that the inability to speak can impact negatively on weaning outcomes. To the investigators' knowledge, this study will be the first to rigorously evaluate, using previously validated measures, the feasibility of the Electrolarynx for establishing communication for mechanically ventilated patients.

Overall Program of Research Hypothesis The investigators hypothesize that restoration of communication using the Electrolarynx can reduce patient anxiety resulting in improvement in weaning outcomes (weaning success and duration) and reduced adverse events associated with inability to communicate such as agitation, delirium, restraint use, and tube/line/device removal. Before being able to test this hypothesis, the feasibility of use of the Electrolarynx needs to be confirmed.

Study Aim The aim of this study is to assess the feasibility of establishing speech with an Electrolarynx for patients receiving ventilation via an endotracheal tube or tracheostomy experiencing difficult weaning and unable to tolerate cuff deflation. Feasibility will be determined in terms of the proportion of participants able to produce intelligible and comprehensible speech as well as ease of, and satisfaction with communication.

ELIGIBILITY:
Inclusion Criteria:

1. endotracheal tube or tracheostomy in situ and unable to tolerate cuff deflation for > one hour
2. alert, awake and able to follow simple commands demonstrated by a Glasgow Coma Score of 15 with the verbal score assigned for the ability to communicate words using non-vocal methods
3. able to read and understand English
4. ≥ 18 years old
5. unimpaired oral-motor capabilities (functional speech structures) assessed by standard oral-peripheral examination by a speech language pathologist and capable of mouthing words in response to orientation questions
6. meets all the above criteria and is anticipated to require mechanical ventilation for a further 5 days
7. consent to participate..

Exclusion Criteria:

1. pre-existing hearing or speech impairment that seriously interferes with communication before hospitalization (as documented in chart or reported by family members)
2. previous diagnosis of dementia identified in the patient's medical history.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Electrolarynx for establishing successful communication defined as the ability to generate speech that is intelligible and comprehensible | Within 5 days of training
  We determined speech intelligibility and comprehensibility using the Assessment of Intelligibility of Dysarthric Speech (AIDS), a validated objective tool for quantifying single-word and sentence intelligibility. Intelligible speech was arbitrarily defined as ≥70% of words identified correctly by raters. Ability to establish comprehensible speech was defined as a difficulty score of ≤ 5 averaged over the five sentences.

SECONDARY OUTCOMES:
Perceived ease and satisfaction with use | Within 5 days of training
  The investigators will use a simplified form of the Ease of Communication scale developed by Menzel that has been adapted and used in studies assessing communication in non-vocal ICU patients. We will use a 5-point Likert type scale to measure satisfaction with 1 indicating very satisfied and 5 indicating not at all satisfied.
Training time | Commencement and completion of training - training is a maximum of five days
  The investigators will record the total time spent to train each participant to use the Electrolarynx
Anxiety | Within 5 days of training
  The investigators will measure anxiety using the Faces Anxiety Scale
Consent rate | One month after completion of study recruitment
  The investigators will document the number of participants that consent and decline
Time to complete research measures | One month after completion of study recruitment
  The investigators will record the time to complete all research procedures
Effectiveness of the Electrolarynx | Within 5 days of training
  The investigators will measure the effectiveness of the Electrolarynx for communication using the Electrolarynx Effectiveness Score

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Toronto East General Hospital, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Care Centre, Toronto, Ontario